CLINICAL TRIAL: NCT02898467
Title: Comparison of Atherothrombosis Markers From Aortic Atheroma in Diabetic and Non-diabetic Patients
Brief Title: Atherothrombosis Markers in Diabetics
Acronym: MADI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Academic Health Science Centres (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/CHU/06
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes; Atherothrombosis; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Thrombosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and serum samples carotid endarterectomy samples urinary samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- diabetics: Type 2 diabetic patients exhibiting fasting glycemia value over 7 mmol/L or glycated hemoglobin value over 6.5% or type 2 diabetic patients under oral anti-diabetic treatment or type 2 diabetic patient under insulin treatment and in which diabetes has been diagnosed after the age of 45 y
  Interventions: Other: diabetics
- non-diabetics: patients without diagnosed diabetes exhibiting fasting glycemia value under 7 mmol/L
  Interventions: Other: non-diabetics

INTERVENTIONS:
Other: diabetics — additional blood and urine collection during usual medical care endarterectomy samples during usual medical care
  Groups: diabetics
Other: non-diabetics — additional blood and urine collection during usual medical care endarterectomy samples during usual medical care
  Groups: non-diabetics

SUMMARY:
Intraplaque hemorrhage is the driving force of atherothrombotic plaque vulnerability to rupture and associated clinical complications. Polymorphonuclear neutrophils (PMNs) represent about 70% of leukocytes and may constitute a source of proteases and oxidants that favour plaque rupture. Our objective is to evaluate PMN activation in atherosclerotic plaque of non-diabetic versus type 2 diabetic patients. For this purpose, investigators will quantify the presence of cell-free DNA, that reflect the formation of neutrophil extracellular traps (NETs) in carotid endarterectomy samples.

DETAILED DESCRIPTION:
Atherothrombotic plaques of type 2 diabetic patients are characterized by increased neovascularization and associated intraplaque hemorrhage relative to non-diabetic patients that could account for a major incidence of clinical complications. In parallel, Type 2 diabetic patients are characterized by an increased intracellular oxidative stress in circulating PMNs leading to a primed phenotype. PMN priming could be triggered via their receptor for advanced glycation endproducts. In particular, glycated albumin may activate NADPH oxidase and thus promote the production of reactive oxygen species. Under strong activation, PMNs have been described to release NETs that are constituted by externalized nucleosomes associating DNA, histones and enzymes initially present in granules (such as myeloperoxidase, matrix metalloproteinase 9 or elastase). Our hypothesis is that in diabetic conditions, PMNs could be activated within atherothrombotic plaques and thus represent a trigger for plaque rupture. In the present study, we will evaluate PMN activation in carotid plaques of diabetic vs non-diabetic patients as well as in plasma samples of the same patients. For this purpose, all patients that will undergo carotid surgery by endarterectomy will be enrolled in our study and blood samples will be collected the day before the surgery for preparation of plasma and serum. The endarterectomy sample will be collected, dissected into culprit area of the plaque (CP) and the adjacent non-complicated plaque (NCP), incubated separately in culture medium for 24h at 37°C. The resulting conditioned medium will be aliquoted and stored at -80°C for the different assessments. A representative section of the CP will be saved at the moment of dissection for histological evaluation (presence of neovessels/intraplaque hemorrhage, calcifications, lipids, etc). Markers of neutrophil activation, of intraplaque hemorrhage, of glycation and of oxidative stress will be quantified in both conditioned medium and plasma.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with planned endarterectomy
* Affiliated to social security rights
* Signed inform consent

Exclusion Criteria:

* pregnancy
* Autoimmune disease, chronic inflammatory disease, neoplasia
* Type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetics and non-diabetics with planned endartectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-11 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Neutrophile activation assessed by free DNA levels in atherothrombotic plaques | On day 1 (day of the surgery)
  Ability of cfDNA concentration in the conditioned medium to discriminate atherothrombotic plaques from diabetic vs non-diabetic patients

SECONDARY OUTCOMES:
Neutrophile activation assessed by other makers than free DNA levels in atherothrombotic plaques | On day 1 (day of the surgery)
  Evaluation of PMN activation by assays other than cfDNA (myeloperoxidase, elastase/antielastase complexes, MMP9/neutrophil-gelatinase associated lipocalin NGAL) in the conditioned media and in plasma
Intraplaque hemorrhage and oxidative stress assessed in plasma and aortic tissue | From day 0 (day before the surgery) to day 1 (day of the surgery)
  Evaluation of markers reflecting the presence of intraplaque hemorrhage and of oxidative stress in conditioned medium and in plasma (CD163, heme, carbonylated proteins, glycated albumin...)
Correlation between plasma and atherothrombotic plaque markers assessement | From day 0 (day before the surgery) to day 1 (day of the surgery)
  Correlations between markers released by the plaque and plasma markers (evaluation of the impact of atherothrombosis at a circulating level)
Atherothrombosis characterization assessed by histological analysis | On day 1 (day of the surgery)
  Histological characterization of plaques assessed by quantification of neovessels, calcification, lipids composition

OTHER OUTCOMES:
Banking of biological samples | From day 0 (day before the surgery) to day 1 (day of the surgery)
  Constitution of a biobank available for different assays of markers and for the discovery of new biomarkers of plaques in type 2 diabetic patients (open approaches, such as differential proteomics)

CONTACTS AND LOCATIONS:
Overall Officials: XAVIER DEBUSSCHE, MD, Principal Investigator — CHU DE LA REUNION
Locations (1):
- Department of endocrinology, University Hospital Reunion Island - Felix Guyon Site, Saint Denis de La Réunion, France

IPD SHARING:
Plan to Share IPD: No